CLINICAL TRIAL: NCT06951659
Title: Clinical, Rehabilitation and Neuroimaging Investigation of Lateropulsion, Graviceptive Neglect and Verticality Perception in Neurosurgical Patients With Brain Tumours: A Prospective Cohort Study
Brief Title: Investigating Visual Verticality Disorder and Lateropulsion in a Neurosurgical Cohort of Patients With Brain Tumours
Status: Recruiting | Type: Observational
Sponsor: The University of Western Australia (Other)
Collaborators: Sir Charles Gairdner Hospital (Other); University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Jimena Garcia-Vega, PhD Candidate, The University of Western Australia
Other Study IDs: RGS5125
Record Dates: First submitted 2025-04-13; First posted 2025-04-30 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-04

CONDITIONS: Brain Tumours
Keywords: Brain tumour; lateropulsion; visual verticality perception; graviceptive neglect; neurosurgery; neuroimaging; structural connectivity; acute care; rehabilitation; neuro-oncology
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with a brain tumour.: This study will investigate a neurosurgical cohort of patients pre and post-brain tumour resection.

SUMMARY:
The overall objective of this research is to investigate the clinical characteristics pre- and post-brain tumour resection with a focus on visual verticality disorder, and lateropulsion, including neuroimaging analysis, of a neurosurgical cohort of patients with brain tumours. This prospective observational cohort study will investigate clinical and neuroimaging characteristics and the relationship between lateropulsion and visual verticality disorder in patients pre- and post-brain tumour resection. Patients (aged 18-80 years, with a confirmed diagnosis of brain tumour and a neurosurgical pathway) will be enrolled from the state-wide Neurosurgery Service of Western Australia at Sir Charles Gairdner Hospital.

DETAILED DESCRIPTION:
Visual verticality perception disorder is the inability to judge the orientation of a vertical line or environment in relation to the Earth's vertical within normal limits, a critical symptom that affects more than half of patients after stroke and impacts global functionality i.e. difficulties maintaining upright posture and stability, poor balance, increased falls risk, and reduced ability to perform daily activities independently. Recently lateropulsion (i.e. a severe postural behavioural expression of visual verticality disorder) has been identified as the primary cause of balance and gait disorders at the subacute stage after stroke. Extending these findings, researchers have reported for the first time that visual verticality disorder and lateropulsion can also be observed in patients with brain tumours in clinical settings. However, there has been no research that has investigated the prevalence and characteristics of visual verticality disorder, and lateropulsion in neurosurgical populations of patients with brain tumours.

This prospective observational study aims to:

1. Describe the relative frequency of lateropulsion and visual verticality disorder pre- and post-surgical resection (up to day 30 post)
2. Compare the visual verticality of patients with and without lateropulsion
3. Investigate the association between lateropulsion and visual verticality disorder post-surgical resection with demographic, clinical and neuroanatomical factors
4. Analyse the predictive factors of functionality, lateropulsion and visual verticality disorder recovery at 30 days post-surgical resection
5. Investigate the factors that influence acute care and rehabilitation LOS
6. Analyse the neural network related to lateropulsion and visual verticality disorder pre- and post-surgical resection.

The preBTR assessments will be completed prior to surgery when possible. In case of an impossibility of assessing preBTR, candidates will be recruited between day 1-5 post-surgery. The postBTR assessments will commence between day 1 to 5 post-surgery (acute postBTR) and comprise of the following clinical variables listed below.

A standardised 'day-30 ± 5 days postBTR (day-30 postBTR) assessment will be performed for all patients either as an inpatient or as an outpatient. All suitable cases assessed during the six-month recruitment period will be reported.

The brain imaging analysis will comprise lesion localisation, lesion volume, indirect structural disconnection-symptom mapping measures (IDSM) and Multivariate Lesion-Symptom Mapping (MLSM).

Abbreviations: preBTR = pre-brain tumour resection, postBTR= post-brain tumour resection

ELIGIBILITY:
Inclusion Criteria:

* Patients of age 18 to 80 admitted to SCGH under the neurosurgery team with a confirmed diagnosis of a brain tumour.
* Only patients who undergo partial or full brain tumour resection and are medically stable.
* Able to provide written informed consent or consent provided by a Research Decision-Maker with the approval of an Independent Medical Practitioner (IMP) as per the Guardianship and Administration Act 1990 (GAA).
* Patients with a support network that enables them to accommodate to travel commitments for assessments if travel to the hospital is required.

Exclusion Criteria:

* Patients who undergo only biopsy will not be included.
* Unable to follow any instructions and complete assessments due to significant medical deterioration.
* Patients who are pregnant.
* Current diagnosis of COVID-19 or respiratory syncytial virus (RSV), or any type of influenza.
* Patients without a support network that enables them to accommodate to travel commitments for assessments if travel to the hospital is required.
* An Advanced Care Health Directive prohibiting decision making by Research Decision-Maker.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the State-Wide Neurosurgical Service of Western Australia (WA) at Sir Charles Gairdner Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2025-12-12 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Visual Verticality Perception (VV, visual graviceptive neglect) | Pre-brain tumour resection, acute post-brain tumour resection (day 1-5), and day 30 post-brain tumour resection (day 30)
  Change in VV: assessment using the bucket test method.
Subjective Haptic Vertical (SHV) test | Pre-brain tumour resection, acute post-brain tumour resection (day 1-5), and day 30 post-brain tumour resection (day 30)
  The SHV test, the participant is blindfolded and asked to align a movable rod or bar to what they perceive as vertical using only their sense of touch (haptic input). This is to isolate somatosensory and vestibular input from visual cues. This will be performed in an upright sitting position to explore graviceptive function and verticality perception.
The Four Point Pusher's Score (4PPS) | Pre-brain tumour resection, acute post-brain tumour resection (day 1-5), and day 30 post-brain tumour resection (day 30)
  The 4PPS is a four-item scale that measures lateropulsion or pusher syndrome. The score for each component is rated on a scale from 0 to 3 (0 to 4 for standing) and the score is based on the severity of resistance or the tilt angle when the patient begins to resist the passive movement. The score for diagnosis of Pusher behaviour is >2 points.
Scale for Contraversive Pushing | Pre-brain tumour resection, acute post-brain tumour resection (day 1-5), and day 30 post-brain tumour resection (day 30)
  A 3-item scale that measures lateropulsion or pusher syndrome, by rating the action / reaction of patients required to keep or change position.
  Scores:
  0= no contraversive pushing
  1. minimum score for each item
  2. maximum score Score on each component >1 indicative of lateropulsion.
Resource Utilisation Group Activities of Daily Living (RUG ADL) | Pre-brain tumour resection, acute post-brain tumour resection (day 1-5), and day 30 post-brain tumour resection (day 30)
  The RUG-ADL score is a 4-item scale measuring motor function with activities of bed mobility, toileting, transfer and eating. The score measures the degree of assistance a patient requires for these activities. The total RUG-ADL score is calculated by summing the scores for the four ADL variables. The total RUG-ADL score ranges from a minimum score of 4 to a maximum score of 18. The higher the score the more assistance the patient requires to complete the four ADL variables.

OTHER OUTCOMES:
Retropulsion | Pre-brain tumour resection, acute post-brain tumour resection (day 1-5), and day 30 post-brain tumour resection (day 30)
  Observed retropulsion of participants in sitting or standing will be documented as 'present' or 'not present'
MD Anderson Symptom Inventory - Brain Tumour (MDASI-BT) | Pre-brain tumour resection, acute post-brain tumour resection (day 1-5), and day 30 post-brain tumour resection (day 30)
  The MDASI-BT is a health-related quality of life questionnaire to assess the severity of symptoms experienced by patients with brain tumours and the interference with daily living caused by these symptoms. The MDASI-BT assesses the severity of symptoms at their worst in the last 24 hours on a 1to 10 numerical scale, with 0 being "not present" and 10 being "as bad as you can imagine", therefore the higher the scores the worst the symptoms and interference. This questionnaire has a total of 28 questions; therefore minimum score is 0 and max 280.
Rehabilitation Complexity Scale - extended version (RCS-E v13) | Pre-brain tumour resection, acute post-brain tumour resection (day 1-5), and day 30 post-brain tumour resection (day 30)
  Rehabilitation Complexity Scale - Extended (RCS-ev13) provides a simple overall measure of resource requirements for rehabilitation including basic care / risk, rehabilitation nursing, therapy (number of disciplines and intensity), medical acuity, equipment needs. The score subscale are divided as follows:
  Care or risk (0-4), Nursing (0-4), Medical (0-4), Therapy (0-8), Equipment (0-2).
  Total score is 22. The higher the score the higher the patient's rehabilitation needs and complexity.
Postural Assessment Scale for Stroke (PASS) | Pre-brain tumour resection, acute post-brain tumour resection (day 1-5), and day 30 post-brain tumour resection (day 30)
  The PASS is an outcome measure specifically designed to assess and monitor postural control after stroke (but also suitable for patients with brain tumours since it is impairment based). It measures the ability of an individual to maintain stable postures and equilibrium during positional changes, using a 4-point scale with a total scoring range from 0 to 36. The PASS consists of 12 items that measure balance in lying, sitting, and standing. The higher the score the more impaired an individual is in regard to maintaining stable postures and equilibrium during positional changes.
Australian Modified Karnofsky Performance Scale (AKPS) | Pre-brain tumour resection, acute post-brain tumour resection (day 1-5), and day 30 post-brain tumour resection (day 30)
  The AKPS is a measure of the patient's functional status or ability to perform their activities of daily living. It is a single score between 10 and 100 assigned by a clinician based on observations of a patient's ability to perform common tasks relating to activity, work, and self-care. The lower the number the more impaired / incapacitated an individual is due to disease progression, and therefore requiring medical assistance or nursing care.
NIH Stroke Scale (NIHSS) | Pre-brain tumour resection, acute post-brain tumour resection (day 1-5), and day 30 post-brain tumour resection (day 30)
  The NIHSS quantifies the impairment caused by a stroke by measuring neurological impairment. this is also commonly used to categorize impairment levels on patients with brain tumours.
  The NIHSS scoring system measures the severity of a stroke (in this case brain tumour neurological impairment), on a scale of 0 to 42. Higher scores indicate greater severity. Stroke severity may be stratified on the basis of NIHSS scores as follows:
  very severe: > 25 severe: 15 - 24 mild to moderately severe: 5 - 14 mild: 1- 5
Montreal Cognitive Assessment (MoCA) | Pre-brain tumour resection and post-brain tumour resection acute (1-5 days)
  Cognitive assessment to determine cognition levels. Normal cognition is defined as a MoCA score of >26 out of 30, mild impairment 18-25 out of 30, severe impairment < 17 out of 30.
Edinburgh Inventory Handedness Assessment | Pre-brain tumour resection
  Questionnaire to assess hand dominance (handedness). It evaluates preference in performing everyday tasks (e.g. writing, throwing, using scissors) using either the left or right hand.
  Scoring: If the preference is for either left or right side, then a "+" is marked on the column for that side. If the preference for a particular side is so strong that one wouldn't use the other side unless forced, then a "++" is marked on that side. If there is no preference for any side, then a "+" is marked on both sides.
  The final score is called the "Laterality Quotient" and is calculated using this formula: laterality quotient = (R-L)/(R+L) x 100
  Handedness is interpreted as follows:
  Left-handedness = less than -40 Ambidexterity = Between -40 and +40 Right-handedness = more than +40
Visual field testing | Pre-brain tumour resection
  Bedside functional visual acuity and visual field testing. Ophthalmology testing results will be used for patients who are incapacitated to complete test.
Nystagmus | Pre-brain tumour resection, acute post-brain tumour resection (day 1-5), and day 30 post-brain tumour resection (day 30)
  Assessment of the presence or absence of nystagmus and semi-spontaneous nystagmus using the Vesticam Binocular IR video goggles with fixation lights (version V2C2C22021) ™
Ocular torsion | Pre-brain tumour resection, acute post-brain tumour resection (day 1-5), and day 30 post-brain tumour resection (day 30)
  Change in ocular torsion: assessment using fundus photography (Phelcom; Eyer device)
Vestibular screening - Benign Paroxysmal Positional Vertigo (BPPV) | Pre-brain tumour resection
  The following assessments with be completed preBTR only. Patients with BPPV report symptoms of vertigo, dizziness, light headedness, and balance problems which can last from seconds to minutes. BPPV will be rated as "positive" or "negative". Positive meaning the patient has a peripheral vestibular dysfunction in the posterior canals.
Spatial neglect | Pre-brain tumour resection, acute post-brain tumour resection (day 1-5), and day 30 post-brain tumour resection (day 30)
  Spatial neglect will be assessed using the conventional Behaviour Inattention Test (BIT), which consists of 6 items: 1) line crossing; 2) letter cancellation; 3)star cancellation; 4) figure and shape copying; 5) line bisection; and 6)representational drawing.
Vestibular screening - Head Impulse Test (HIT) | Pre-brain tumour resection
  The following assessments with be completed preBTR only. The HIT is a clinical assessment technique used to evaluate the vestibular ocular reflex (VOR), which helps maintain stable vision during head movements.
  the evaluation of the HIT will be as either "present" or "not present" and the notation if there are corrective saccades with head movement to either "right" or "left".
Brain magnetic resonance imaging (MRI) | Pre-brain tumour resection, and day 30 post-brain tumour resection (day 30)
  The structural integrity of the visual verticality and lateropulsion network will be evaluated using diffusion MRI i.e. Lesion localisation, lesion volume, indirect structural disconnection-symptom mapping measures (ISDSM) i.e. tract disconnection, parcel disconnection.
Vestibular screening - Head Shake test | Pre-brain tumour resection
  The following assessments with be completed preBTR only. The head shake test is a diagnostic tool used to evaluate balance disorders, dizziness, and vertigo. During the test the clinician rapidly shakes the patient's head to elicit nystagmus, with can indicate vestibular system issues. Documentation will be as either "present" or "not present" and the notation if there is nystagmus present (corrective saccades) after 30 seconds of head shaking.

CONTACTS AND LOCATIONS:
Overall Officials: Taiza GS Edwards, PhD, Principal Investigator — The University of Western Australia; Anne-Marie Hill, PhD, Principal Investigator — The University of Western Australia
Locations (1):
- Sir Charles Gairdner Osborne Park Health Care Group, Perth, Western Australia, Australia

IPD SHARING:
Plan to Share IPD: Undecided